CLINICAL TRIAL: NCT05316857
Title: A Phase I, Single-center, Open-label, Fixed-sequence Clinical Study to Evaluate the Effects of Multiple Administrations of Rifampin or Itraconazole on the Pharmacokinetic Characteristics of a Single Administration of Orelabrutinib Tablets in Healthy Subjects
Brief Title: DDI Study of Orelabrutinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ICP-CL-00117
Record Dates: First submitted 2022-03-25; First posted 2022-04-07 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Healthy Person
MeSH Terms: interventions — orelabrutinib; Rifampin; Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orelabrutinib + Rifampin (Other): Orelabrutinib is a white, round, uncoated table,Subjects take high dose orelabrutinib in the first day and the tenth day.
  Rifampin is a capsule,Subjects take 600mg QD rifampin in the third day to the eleventh.
  Interventions: Drug: Orelabrutinib + Rifampin
- Orelabrutinib + Itraconazole (Other): Orelabrutinib is a white, round, uncoated table,Subjects take low dose orelabrutinib in the first day and the eighth day.
  Itraconazole is a capsule,Subjects take 600mg QD rifampin in the third day to the tenth.
  Interventions: Drug: Orelabrutinib + Itraconazole

INTERVENTIONS:
Drug: Orelabrutinib + Rifampin — Orelabrutinib + Rifampin
  Arms: Orelabrutinib + Rifampin
Drug: Orelabrutinib + Itraconazole — Orelabrutinib + Itraconazole
  Arms: Orelabrutinib + Itraconazole

SUMMARY:
This is a phase I, single-center, open-label, fixed-sequence clinical study. The primary objective was to evaluate the effects of multiple administrations of rifampin or itraconazole on the pharmacokinetic characteristics of a single administration of orelabrutinib tablets in healthy Chinese subjects. The secondary objective was to evaluate the safety and tolerability of rifampicin or itraconazole combined with orelabrutinib tablets in healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who can fully understand the objectives, nature, methods and possible adverse reactions of the trial, and volunteers to be the subject, and has signed an informed consent form before the start of any study procedure, and guarantees that any procedure will be participated in by himself/herself;
2. Male or female subjects aged between 18 and 45 years old (inclusive) at the time of screening;
3. Body weight ≥50 kg for male subjects, ≥45 kg for female subjects, and a body mass index (BMI) of 19 to 26.0 kg/m2 (inclusive);
4. Be able to communicate well with investigator, and understand and comply with the requirements of this study.

Exclusion Criteria:

1. Complete physical examination, routine laboratory tests, cardiac color ultrasound and other examinations are abnormal with clinical significance;
2. Hepatitis B surface antigen or E antigen, hepatitis C antibody, human immunodeficiency virus (HIV) antibody, or syphilis antibody are positive;
3. C-reactive protein for novel coronavirus screening is abnormal with clinical significance, or the novel coronavirus nucleic acid testing is positive;
4. Have received any drugs and therapy which are in the study protocol within 1 month before screening
5. Have taken prescription drugs, over-the-counter drugs, dietary supplements, or Chinese herbal medicine within 14 days before the first administration of the investigational drug
6. Have any history of clinically serious diseases, or diseases or conditions that the investigator believes may affect the results of the study.
7. Subject who has a childbirth plan during the study period and within 3 months after the end of the study, or the subject and his/her partner do not agree to take strict contraceptive measures during this period;
8. Other subjects judged by the investigator as unsuitable to participate in this study NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 3 months
  To preliminarily obtain pharmacokinetic (PK) data of Orelabrutinib in the treatment of advanced solid tumors include the peak plasma concentration (Cmax)

SECONDARY OUTCOMES:
Tmax | up to 3 months
  To preliminarily obtain pharmacokinetic (PK) data of Orelabrutinib in the treatment of advanced solid tumors include Time to Maximum Plasma Concentration(Tmax)
Incidence of Treatment-Emergent Adverse Events | up to 3 months
  To evaluate the safety and tolerability of Orelabrutinib

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China